CLINICAL TRIAL: NCT07170891
Title: Effects of Inspiratory Muscle Training Combined With Circadian Rhythm-based Running Programs in Children Male Football Players
Acronym: Circadian IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, ASSOC. PROF., Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E-95674917-108.99-282503
Record Dates: First submitted 2025-06-20; First posted 2025-09-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: 10-13 Age; Inspiratory Muscle Training; Running; Circadian Rhythm
Keywords: football players; exercise; agility; running training; circadian rhythm; inspiratory muscle training; performance; Children
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: In this study, a parallel two-group pre-test-post-test randomized controlled trial was conducted according to CONSORT guidelines [14]. All participants and their parents were given detailed information about the study before it commenced, and written informed consent was obtained in accordance with the ethical principles described in the Declaration of Helsinki. Help was received from a third-level athletics coach for planning and implementing running exercises to be used in the project. The aim of this study is to investigate the effects of additional inspiratory muscle training (IMT) on exercise tolerance, agility performance, and respiratory parameters in 10-12-year-old male football players who have been training regularly for at least two years, based on their chronotype. G*Power 3.1 to determine the sample size of the study. Based on this analysis, it was determined that a minimum of 20 participants per group was required
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (Active Comparator): no exercise group
  Interventions: Other: Control
- MORNİNG RUNNİNG+IMT (Active Comparator): Inspiratory muscle training was performed in addition to morning running
  Interventions: Device: Morning Running and IMT
- EVENİNG RUNİNG+IMT (Active Comparator): Inspiratory muscle training was performed in addition to evening running
  Interventions: Device: Inspiratory muscle training and evening running

INTERVENTIONS:
Device: Morning Running and IMT — Inspiratory muscle training was performed in addition to morning running
  Arms: MORNİNG RUNNİNG+IMT
Device: Inspiratory muscle training and evening running — Inspiratory muscle training was performed in addition to evening running
  Arms: EVENİNG RUNİNG+IMT
Other: Control — non-exercise group
  Arms: CONTROL

SUMMARY:
In this study, a parallel two-group pre-test-post-test randomized controlled trial was conducted according to CONSORT guidelines. All participants and their parents were given detailed information about the study before it commenced, and written informed consent was obtained in accordance with the ethical principles described in the Declaration of Helsinki. Help was received from a third-level athletics coach for planning and implementing running exercises to be used in the project. The study was designed according to the rules of the Declaration of Helsinki and approved by the ethics committee for scientific research of Gümüşhane University (at its meeting on 20.09.2024 and number 2024/7; decision number E-95674917-108.99-282503). The aim of this study is to investigate the effects of additional inspiratory muscle training (IMT) on exercise tolerance, agility performance, and respiratory parameters in 10-12-year-old male football players who have been training regularly for at least two years, based on their chronotype. A power analysis was conducted using G*Power 3.1 to determine the sample size of the study. The effect size (d) was found to be 1.12 (α = 0.05, 1-β = 0.95, η²p = 0.8). Based on this analysis, it was determined that a minimum of 20 participants per group was required. However, to mitigate potential issues, it was decided to include 25 participants, an additional 25%, in each group.

Participants visited the laboratory three times. During the first visit, the familiarization procedure was performed; participants were administered the Morningness-Eveningness Scale for Children questionnaire and divided into 3 groups according to the results. Then, pulmonary function tests (PFT), maximum inspiratory pressure (MIP), expiratory pressure (MEP), six-minute walk test (6MWT), inspiratory muscle training (IMT), and running training procedures were applied. In the second visit, PFT and MIP-MEP tests, agility and 6MWT tests were performed and their performances were recorded. After the six-week training period, participants' final measurements were taken at the third and final visit. Subsequent to the completion of the six-week training period, the participants' final measurements were obtained during the final visit. The experimental trials were conducted at a consistent time each day, between 9:00 and 12:00. Prior to the commencement of the trials, participants were instructed to abstain from high-intensity physical activity.

The inclusion criteria were as follows: a) Candidates must have at least two years of active football training, b) be between the ages of 10 and 13, c) be in good general health, d) have no known respiratory or cardiovascular conditions, e) provide written informed parental consent. The following criteria were used to determine exclusion from the study: The subject's medical history includes the following: a) A history of lung disease or a current upper respiratory tract infection, b) A history of current injury, c) Medication use that may affect breathing or performance, d)Individuals with FEV1/FVC<70 e) Participation in similar studies within the last six months

DETAILED DESCRIPTION:
Body composition measurement The height of the participants was measured using a standard height meter (Seca 769, Seca, Hamburg, Germany) with an accuracy of 0.1 centimeter while leaning against a wall without shoes. Body weight was measured using a digital scale (Beurer, model GS27) with an accuracy of 0.1 kilograms before and after the IMT program, which was itself incorporated into the 6-week running program. The participants' body weight was measured in kilograms (kg) without shoes and wearing shorts and a T-shirt to avoid affecting the results.

The Morningness-Eveningness Scale for Children (MESC) The Morningness-Eveningness Scale for Children (MESC), developed by Carskadon et al. (1993), is a tool designed to assess the daily preferences of school-age children. The scale under consideration consists of 10 items with four or five response options. Scores on the scale range from 10 to 43. Established 21 and 35 as the cut-off points for the scale. A positive correlation has been demonstrated between children's preference for mornings and their score on the scale. That is to say, as the score on the scale increases, the preference for mornings concomitantly increases. Scores ranging from 22 to 34 points are indicative of an intermediate type, while scores of 21 or below are associated with an evening type. Scores of 35 points and above are considered to indicate a morning type. The validity and reliability of the Turkish version of the scale were previously examined by Önder and Beşoluk (2013), who determined a Cronbach's alpha value of 0.72. In the context of the study, subjects who attained scores below 21 points were allocated to the evening group. Those who scored between 22 and 34 points were designated as the control group, which comprised individuals who engaged exclusively in jogging. Subjects who scored 35 points and above were assigned to the morning group.

505 Agility test This test consists of measuring the time taken to complete the last 5 meters of a 15-meter track. The time within the first 10 m from the start of the test is not included in the test score. When the next 5 m distance is passed for the first time, the recording begins and stops when the same distance is covered in return.

Six-Minute Walk Test (6MWT) Protocol The 6MWD test is a reliable and valid functional test that can be used to assess exercise tolerance and endurance in healthy children. The rationale behind our selection of this particular evaluation method stems from its status as the most pragmatic and ergonomic approach to appraising the submaximal extent of functional exercise capacity. The Six Minute Walk Test (6MWT) instructions were provided to all participants by an exercise physiologist. The participants were instructed to walk as fast as possible while maintaining a comfortable pace for the duration of six minutes along a pre-measured straight path. During the test, the assessor recorded the time and provided standardized encouragement at each minute interval. The assessor also tallied the number of laps completed by each participant. At the sixth minute, the participants halted at their position on the path, and the assessor recorded the total distance traversed for the final lap. The evaluator then calculated and recorded the total distance walked over the 6-minute period.

Pulmonary function tests FEV1, FEV1/FVC (Tiffenau index), and FVC capacity were analyzed via a CPFS/D USB spirometer from MGF Diagnostics (Saint Paul, Minnesota, USA). Measurements were taken between 15:00 and 17:00 for all participants to obtain the highest spirometric throughput. Participants with FEV1/FVC <75%, any chronic or pulmonary disease, medication that could affect lung function, or a history of upper respiratory tract infection were excluded from the study. Lung function tests were performed with the partic-ipants in the standing position. During the tests, the participants wore a nose clip and were instructed to hold their lips tightly around the mouthpiece to prevent air from escaping.

Respiratory muscle strength Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) were measured via a hand-held portable oral pressure meter (MicroRPM, CareFusion Micro Medical, Kent, UK) according to the American Thoracic Society and European Respiratory Society guidelines. With the appropriate filters and holders in place, the nasal airway was closed with a clip. The mouthpiece assembly included a 1 mm hole to prevent glottic closure and minimize the contribution of the buccinator muscles during inspiration. Inspiratory and expiratory maneuvers were performed in the standing position, with MIP and MEP measurements starting at the residual volume and total lung capacity, respectively, and continuing for at least 1 second. The measurements were repeated until there was a 5% difference between the two best results, and the results were recorded as the mean cm H2O.

Running training The morning running sessions were performed between 08:00 and 10:00, the evening sessions were performed between 18:00 and 20:00, and the control group, which only jogged, performed their sessions between 12:00 and 15:00. The exercise intensity for each participant in the running groups was determined as 50% of their heart rate (HR) calculated using the Karvonen formula: Target HR = [(220 - age - rest HR) × intensity] + rest HR. HR was monitored from the first week of training using a telemetric heart rate monitor (Polar M400, Finland). As environmental conditions can affect airway epithelial responses during high-intensity exercise, all participants performed continuous running exercises on a soccer field in Kelkit, Gümüşhane, Turkey (altitude: 1373m). Each session lasted 50 minutes, including a 10-minute warm-up and cool-down each, and was performed at the set target HR three days per week over a six-week period. All sessions were supervised by trained coaches. Warm-up and cool-down routines included static stretching and light exercises targeting relevant muscle groups. Coaches were responsible for monitoring athletes' running technique and speed, ensuring safety and providing motivation. Both groups were adequately hydrated throughout the sessions to prevent dehydration.

Inspiratory muscle training (IMT) Inspiratory muscle training (IMT) was performed using the POWERbreathe® device (POWER® Breathe Classic, IMT Technologies Ltd., Birmingham, UK). The IMT protocol was administered twice daily, in the morning and evening, for a period of six weeks, with the intervention occurring five days per week. Each training session comprised 30 breathing cycles (totaling 60 breathing cycles per day), and participants performed these exercises separately in the morning and evening. Prior to the administration of the POWERbreathe® device, the resistance setting was calibrated to 40% of the participant's maximum inspiratory pressure (MIP), as reported in the study by Çelikel et al. (2025). The initial MIP value was increased by 10% on a weekly basis. The training sessions were overseen by a certified trainer, who ensured that participants adhered to proper form. The morning IMT sessions were held between 8:00 and 10:00, and the evening sessions were held between 17:00 and 20:00.

Statistical analysis The research data were analyzed via IBM SPSS Statistics 24. Descriptive data are presented as the means and standard deviations. The normality of the data was examined via the Kolmogorov-Smirnov test, which revealed that the data were normally distributed. For parametric data, the dependent group t test (paired samples t test) was used for within-group, pretest, and posttest comparisons, and ANOVA was used for the developmental results obtained using the posttest-pretest difference formula. In addi-tion, in the comparison of paired groups, the effect size was calculated according to Cohen's d formula ((M2 - M1) ⁄ the pooled standard deviation). Moreover, it was interpreted as follows: 0 - 0.19 insignificant, 0.20 - 0.59 small, 0.6 - 1.19 moderate, 1.20 - 1.99 large, and ≥ 2.00 very large. Statistical significance was based on a p value of < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must have at least two years of active football training
* be between the ages of 10 and 13,
* be in good general health
* have no known respiratory or cardiovascular conditions,
* provide written informed parental consent.

Exclusion Criteria:

* A history of lung disease or a current upper respiratory tract infection,
* A history of current injury,
* Medication use that may affect breathing or performance,
* Individuals with FEV1/FVC<70
* Participation in similar studies within the last six months

Ages: 10 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Agility (505 Agility Test) | 8 weeks.
  Agility (505 Agility Test): Change from baseline to 8 weeks.
6-Minute Walk Test (6MWT) | 8 weeks.
  6-Minute Walk Test (6MWT): Change from baseline to 8 weeks.

SECONDARY OUTCOMES:
Respiratory Muscle Strength | 8 weeks.
  Maximal Expiratory Pressure (MEP) Maximal Inspiratory Pressure (MIP) Description: Maximal Inspiratory Pressure (MIP): Change from baseline to 8 weeks. Time Frame: 8 weeks.
Pulmonary Function | 8 weeks.
  Pulmonary Function (FEV1, FVC, FEV1/FVC): Change from baseline to 8 weeks. Respiratory Parameters
  -Pulmonary Function Tests (PFT): FEV1 (Forced Expiratory Volume in 1 second) FVC (Forced Vital Capacity) FEV1/FVC ratio (Tiffenau index)

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane Univetsity, Kelkit, Gümüşhane Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE PERSONAL DATA WILL BE SHARED IF REQUESTED.